CLINICAL TRIAL: NCT00836186
Title: Cytokine Expression During Radiation for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J08130; NA_00024399 (Other: JHM IRB)
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer
Keywords: Cytokine; Tumor Marker; Disparities
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: This is a prospective study designed to analyze tumor markers and pathologic data in order to examine the prediction of tumor response to radiation therapy.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation therapy (Other): Women with non-metastatic breast cancer status post lumpectomy to negative margins and who are receiving whole breast irradiation as per standard treatment plan.
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy — Patients will receive whole breast radiation therapy at a dose of 180-200 centigray (cGy) per fraction for 23-27 fractions to a total dose of 4600 - 4860 cGy. Additional radiation to the lumpectomy bed (Boost) is at the discretion of the treating physician. The total dose to the tumor bed cannot exceed 6600 cGy.

SUMMARY:
To assess the magnitude and frequency of changes in chemo/cytokine expression in women receiving radiation treatment. To asses the impact of race/ethnicity on the magnitude and frequency of changes in chemo/cytokine expression during radiation therapy for breast cancer. And finally to assess the interaction between radiation-induced chemo/cytokine expression changes, and race/ethnicity, with respect to normal tissue reactions to radiation and tumor-associated outcomes.

DETAILED DESCRIPTION:
It is well recognized that the diagnostic and therapeutic gains made in the management of breast cancer over the last 2 decades are not fully realized by all groups. African American women with breast cancer have greater risk of recurrence, shorter overall survival, shorter survival after relapse, worse toxicity and worse cosmetic outcome than their Caucasian counterparts. These differences in outcome persist even when controlling for age, and stage at presentation. Being similarly treated with modern breast conserving therapy (lumpectomy and adjuvant whole breast irradiation) at recognized centers of excellence does little to alleviate the disparities in outcomes. Controlling for socioeconomic factors decreases the severity of these disparities, but it does not completely explain them. Theories abound as to the cause of outcome inequality. Many of these theories take either a psychosocial, or biologic bent. One potential biologic cause may be chemokine and cytokine expression.

Chemokines and cytokines (chemo/cytokines) are proteins and peptides used for cell signaling. Primarily secreted by T cells and macrophages, they influence cellular activation, differentiation, and function and act as mediators for inflammatory and immune responses. There has been substantial research linking some of these chemo/cytokines [Tumor necrosis factor alpha (TNFα), platelet derived growth factor (PDGF), Transforming growth factor beta (TGFβ), interleukin (IL)-6,and IL-8] to tumor promotion and progression. For example, TNFα has been linked to greater cell survival despite genomic injury which in turn leads to greater genetic alterations and malignant transformation. TNFα has been associated with breast cancer progression and metastases. Blocking the receptor for PDGF appears to decrease the metastatic potential of breast cancer cell lines. TGFβ inhibits T cell and B cell lymphocytes and natural killer cell cytotoxicity. This immuno-suppression has been shown to promote tumor progression in mammary cancer cells lines. The ability of TGFβ to promote tumor progression is so well recognized that it has become a therapeutic target by some researchers. Interferon gamma (IFNγ) has been shown to inhibit mammary cancer cell proliferation and angiogenesis in vitro and in vivo. Clinically, Lyon et al reported significantly higher circulating levels of TNFα, IL-6, and IL-8 in women with breast cancer compared to women with a negative breast biopsy. Additionally, researchers have directly correlated increased levels of IL-6 with the development and progression of breast cancer, and decreased overall survival (OAS). Conclusion: Expression of certain chemokines and cytokines is associated with development and progression of breast cancer.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patient must be 18 years of age or older
* Patients must have histologically confirmed (by routine H&E staining) adenocarcinoma of the breast any T, any N, M0 disease
* Patients must have undergone a segmental mastectomy (SM) with a level I and ll axillary dissection or sentinel lymph node biopsy. Surgical margins at time of local surgery must be negative greater or equal to 2mm for both invasive carcinoma and for non-invasive ductal carcinoma Patients who have post-operative margins which are negative but less than 2mm will be considered eligible if the surgeon states that the margin in question cannot be improved.
* Patients must be registered such that radiation therapy begins within 10 weeks of last surgery
* Patients must have a performance status 0 or 1 by Eastern Cooperative Oncology Group (ECOG) criteria or a 80-100 Karnofsky Performance Scale at time of consult
* Women of all races and ethnic groups are eligible for this trial

EXCLUSION CRITERIA:

* Patients must not have received prior radiation therapy to the breast at any time for any reason
* Patients with squamous carcinomas or sarcomas of the breast cancer are not eligible
* Patients treated with a mastectomy are NOT eligible
* Any patient with active local-regional disease prior to registration is not eligible
* No other prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or any other cancer from which the patient has been disease-free for at least 5 years
* Patients must not be pregnant due to the potential for fetal harm as a result of this treatment regimen. Women of child-bearing potential must use effective non hormonal contraception while undergoing radiation therapy
* Patients must not have a serious medical or psychiatric illness which prevents informed consent or compliance with treatment

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-11-13 (Actual); Primary Completion 2014-11-26 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Wright, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - The Johns Hopkins University School of Medicne, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiation Therapy: Women with any non-metastatic breast cancer status post lumpectomy to negative margins and who are receiving whole breast irradiation as per standard treatment plan.
  Radiation therapy: Patients will receive whole breast radiation therapy at a dose of 180-200 centigray (cGy) per fraction for 23-27 fractions to a total dose of 4600 - 4860 cGy. Additional radiation to the lumpectomy bed (Boost) is at the discretion of the treating physician. The total dose to the tumor bed cannot exceed 6600 cGy.
Period: Overall Study
Arm/Group | Radiation Therapy
Started | 82
Completed | 81
Not Completed | 1
Not completed — Blood could not be drawn | 1

BASELINE CHARACTERISTICS:
Groups:
- Radiation Therapy: Women with any non-metastatic breast cancer status post lumpectomy to negative margins and who are receiving whole breast irradiation as per standard treatment plan.
  Radiation therapy: Patients will receive whole breast radiation therapy at a dose of 180-200 cGy per fraction for 23-27 fractions to a total dose of 4600 - 4860 cGy. Additional radiation to the lumpectomy bed (Boost) is at the discretion of the treating physician. The total dose to the tumor bed cannot exceed 6600 cGy.
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 66
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 41
  White | 38
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 81
  Canada | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Proteins Expressed Differently in Response to Receiving Radiation Therapy
Description: Number of proteins that are expressed differently in response to receiving radiation therapy for breast cancer. The data reflect the total number of proteins pooled across all participants.
Time Frame: 2 - 4 weeks post radiation therapy
Population: Analysis of blood samples were completed on 65 patients and therefore data was only available for these 65 participants.
Measure: Number; unit: Proteins
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 65
Proteins | 31

2. Secondary Outcome: Number of Proteins With Differential Expression by Race/Ethnicity
Description: To asses the impact of race/ethnicity on the expression of proteins after radiation therapy for breast cancer. The data reflect the total number of proteins pooled across all participants.
Time Frame: 2 - 4 weeks post radiation therapy
Population: Analysis of blood samples were completed on 65 patients and therefore data was only available for these 65 participants.
Measure: Number; unit: Proteins
Groups:
- Radiation Therapy: Women with non-metastatic breast cancer status post lumpectomy to negative margins and who are receiving whole breast irradiation as per standard treatment plan.
  Radiation therapy: Patients will receive whole breast radiation therapy at a dose of 180-200 cGy per fraction for 23-27 fractions to a total dose of 4600 - 4860 cGy. Additional radiation to the lumpectomy bed (Boost) is at the discretion of the treating physician. The total dose to the tumor bed cannot exceed 6600 cGy.
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 65
Proteins | 4

3. Secondary Outcome: Number of Metabolites That Changed Differentially on the Basis of Patient Toxicity
Description: The chemo/cytokine expression changes with respect to radiation toxicities as assessed by number of metabolites that changed differentially on the basis of patient toxicity. The data reflect the total number of metabolites pooled across all participants.
Time Frame: 2 - 4 weeks post radiation therapy
Population: Analysis of blood samples were completed on 65 patients and therefore data was only available for these 65 participants.
Measure: Number; unit: metabolites
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 65
metabolites | 39

ADVERSE EVENTS:
Description: Adverse Event data was not collected.
Arm/Group | Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No